CLINICAL TRIAL: NCT07119697
Title: Efficacy of Shacklock Neural Mobilization vs. McKenzie Extension Principle in Lumbar Radiculopathy: A Randomized Comparative Trial on Pain and Functional Disability
Brief Title: Shacklock Neural Mobilization vs. McKenzie on Pain and Functional Disability in Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2021-10
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Radiculopathy
Keywords: Oswestry Disability Index (ODI); McKenzie Method; Neural Mobilization; Radiculopathy; Exercise Therapy; Rehabilitation Outcome
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNM Group (Experimental): SNM Group exhibited 22 participants who received allocated intervention, including Shacklock Neural Mobilization and hydrocollator packs for 15-20 minutes per session, 3-5 days weekly for three weeks.
  Interventions: Other: Shacklock Neural Mobilization; Other: Hydrocollator hot packs
- MEP Group (Active Comparator): MEP Group exhibited 22 participants who received allocated intervention, including the McKenzie Extension Principle and hydrocollator packs for 15-20 minutes per session, 3-5 days weekly for three weeks.
  Interventions: Other: McKenzie Extension Principle; Other: Hydrocollator hot packs

INTERVENTIONS:
Other: Shacklock Neural Mobilization — In the SNM group, participants lay supine with hips neutral and knees flexed to 45 degrees. Therapists applied the remote slider technique by extending the knee near end-range and dorsiflexing the ankle to 15 degrees, performed in 3 sets of 15 reps with 30-second rests. Each session lasted 20 minutes including setup. Progression was made by increasing hip flexion in 5 degrees increments when a VAS pain reduction of ≥2 cm was observed. This technique, based on neurodynamic principles, was designed to reduce neural mechanosensitivity and improve mobility in patients with lumbar radiculopathy.
  Arms: SNM Group
Other: McKenzie Extension Principle — MEP group was treated with MEP in a prone position, starting with 10 repetitions of active trunk extension, holding end-range for 3 seconds. If no symptom centralization occurred, therapists progressed from patient-applied overpressure (EIL-POP) to clinician-applied grade III mobilizations (3 oscillations/second), following McKenzie's force progression model. Each session included 3 sets of 10 repetitions with 1-minute rest between sets, totaling 15 minutes of active intervention. For unilateral symptoms, the approach advanced to hips-off-center techniques involving a 15 degree lateral shift. This graded sequence aimed to reduce nerve root compression and promote symptom centralization.
  Arms: MEP Group
Other: Hydrocollator hot packs — Both groups received standardized thermotherapy using hydrocollator-heated moist hot packs (40 degrees centigrade, wrapped in 6-8 towel layers) applied to the lumbar region for 15-20 minutes to improve tissue compliance and reduce pain. Participants were positioned prone or side-lying based on comfort and symptom severity; semi-prone positions with pillow support were used for those with heightened sensitivity to maintain spinal neutrality. Thermotherapy was administered five times in week 1 and three times weekly during weeks 2-3. Skin condition and comfort were monitored. This pre-treatment method promoted transient pain relief and muscle relaxation, enhancing tolerance to subsequent therapeutic interventions.

SUMMARY:
This randomized comparative trial evaluates the efficacy of Shacklock neural mobilization versus the McKenzie extension principle in patients with lumbar radiculopathy. The study aims to compare both interventions in terms of their effectiveness in reducing pain and improving functional disability. Outcomes will be measured using validated tools such as the Visual Analog Scale (VAS) for pain and the Oswestry Disability Index (ODI). The trial seeks to inform evidence-based physiotherapeutic approaches for managing lumbar radiculopathy.

DETAILED DESCRIPTION:
This randomized comparative trial is designed to assess and compare the efficacy of Shacklock Neural Mobilization (SNM) and the McKenzie Extension Principle (MEP) in the management of lumbar radiculopathy. Lumbar radiculopathy is commonly associated with nerve root compression, resulting in significant pain and functional limitations. While SNM focuses on restoring normal neurodynamic mobility and reducing mechanosensitivity of the nervous system, MEP targets spinal mechanical derangements through repeated extension movements. Despite their widespread clinical use, direct comparative evidence on their effectiveness remains limited.

The study utilizes a two-arm, parallel-group design with repeated measures. Participants diagnosed with lumbar radiculopathy were randomly assigned to one of two intervention groups: the SNM group or the MEP group. Each group received their respective intervention over a structured three-week treatment period.

Interventions were administered by qualified physiotherapists following standardized protocols. Pain intensity and functional disability were measured using the Visual Analog Scale (VAS) and the Oswestry Disability Index (ODI), respectively. Assessments were conducted at baseline and weekly thereafter until the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

It required participants to have subacute lumbar radiculopathy (3-6 months duration) with radiating pain to or beyond the knee, with or without neurological signs, and MRI-confirmed mild disc bulge. Eligibility also required meeting at least three of four standardized test item cluster criteria and the ability to read and understand English.

Exclusion Criteria:

It included a history of spinal trauma or surgery, presence of systemic diseases (such as rheumatoid arthritis or diabetes), severe disc pathology (e.g., sequestration), spinal deformities (e.g., scoliosis >10°), chronic radiculopathy lasting more than one year, or current use of nonsteroidal anti-inflammatory drugs (NSAIDs).

Ages: 25 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 3 weeks
  Pain intensity was measured using the Visual Analog Scale (VAS), a 10-cm horizontal line anchored by no pain (0) and worst imaginable pain. The VAS is a validated and reliable tool, with excellent test-retest reliability (ICC = 0.94) and strong correlations with other pain measures. Patients marked their pain after a 10-minute rest to minimize activity-induced fluctuations, and assessments were conducted at standardized time points throughout the intervention period.
Functional Disability | 3 weeks
  The Oswestry Disability Index (ODI) version 2.1a was used to assess functional limitations related to lumbar radiculopathy. This 10-item questionnaire, scored from 0 to 100%, has demonstrated excellent internal consistency (α = 0.90) and test-retest reliability (ICC = 0.91) in lumbar spine conditions. Participants completed the ODI independently under standardized conditions, ensuring accurate assessment of daily activity limitations associated with radiculopathy.
Lumbar Range of Motion | 3 weeks
  Spinal mobility was objectively assessed using a modified Schober's test combined with digital inclinometry (Baseline® inclinometer). Flexion was measured using Schober's method, while extension was assessed with the inclinometer placed at the T12-L1 level. Three consecutive readings were taken and averaged for each direction following a standardized warm-up protocol to minimize viscoelastic tissue effects and ensure consistency across assessments.
Neurodynamic Assessment | 3 weeks
  The Straight Leg Raise (SLR) test was conducted using a standardized protocol known for high sensitivity in detecting nerve root compression when combined with ankle dorsiflexion. A Baseline® 12 plastic goniometer was used to measure the angle at which radicular symptoms were first reproduced. The hip was moved at a controlled rate of 10 degree, second to differentiate neural from musculoskeletal responses. This approach allows for consistent and reliable monitoring of neurodynamic changes throughout the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ahmad H. Alghadir, PhD, Study Chair — Rehabilitation Reseach Chair; King Saud University
Locations (1):
- King Saud University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Study title, brief and descriptive summary, Methodology, including, Study design, setting, Study protocol, outcomes, iterventions may be shared.
Supporting Information: Study Protocol
Time Frame: 6 weeks
Access Criteria: Peer reviewing intended